CLINICAL TRIAL: NCT00866541
Title: Flow Proportional Pressure Support as a New Mode of Spontaneous Breathing Assist - Evaluation of Objective and Subjective Measured Data in Volunteers
Brief Title: Flow Proportional Pressure Support in Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Dr. med. Daniel Steinmann, University Medical Center Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 327/07
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: resistance; flow proportional pressure support; pressure support ventilation; volunteers; assistant breathing; breathing comfort and objective breathing data

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- volunteers (Experimental): artificial increased respiratory resistance
  Interventions: Device: artificial increased resistance (flow proportional pressure support)

INTERVENTIONS:
Device: artificial increased resistance (flow proportional pressure support) — respiratory resistance is increased by interpose of an artificial resistance tool in the in- and expiratory airways of the mechanical respirator

SUMMARY:
Flow proportional pressure support (FPPS) is a new mode of spontaneous breathing assistance. In patients with increased respiratory resistance the role of FPPS in comparison with the pressure support assist breathing mode is still unclear. In this study the investigators evaluate objective and subjective measured data in healthy volunteers with artificial increased resistance and FPPS breathing assistance.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* ASA I and II

Exclusion Criteria:

* refusal of written informed consent
* chronic respiratory or cardiac diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
pressure support | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinmann, MD, Principal Investigator — University Medical Center Freiburg
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Background] Mols G, Vetter T, Haberthur C, Geiger K, Guttmann J. Breathing pattern and perception at different levels of volume assist and pressure support in volunteers. Crit Care Med. 2001 May;29(5):982-8. doi: 10.1097/00003246-200105000-00018. PMID 11378608
- [Background] Mols G, von Ungern-Sternberg B, Rohr E, Haberthur C, Geiger K, Guttmann J. Respiratory comfort and breathing pattern during volume proportional assist ventilation and pressure support ventilation: a study on volunteers with artificially reduced compliance. Crit Care Med. 2000 Jun;28(6):1940-6. doi: 10.1097/00003246-200006000-00042. PMID 10890645
- [Background] Mols G, Rohr E, Benzing A, Haberthur C, Geiger K, Guttmann J. Breathing pattern associated with respiratory comfort during automatic tube compensation and pressure support ventilation in normal subjects. Acta Anaesthesiol Scand. 2000 Mar;44(3):223-30. doi: 10.1034/j.1399-6576.2000.440302.x. PMID 10714832
- [Background] Guttmann J, Bernhard H, Mols G, Benzing A, Hofmann P, Haberthur C, Zappe D, Fabry B, Geiger K. Respiratory comfort of automatic tube compensation and inspiratory pressure support in conscious humans. Intensive Care Med. 1997 Nov;23(11):1119-24. doi: 10.1007/s001340050467. PMID 9434916